CLINICAL TRIAL: NCT03009994
Title: Exteriorization Versus Non-exteriorization of the Uterus During Repair of Uterine Incision in a Repeated Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Prof, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EUR
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Intrapartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exteriorization group (Other): After delivery of the fetus and placenta, the surgeon bring uterus yet out from peritoneal cavity by manual handling of the uterus uterus from fundus and extracted out of the abdominal cavity before starting to close it. After repair of the uterus , uterus returned to abdominal cavity and repair anterior abdominal wall as following.
  Interventions: Procedure: Repair of uterine incision; Procedure: Exteriorization of the uterus
- Non exteriorization group (Other): Uterine incision will be repaired intra abdominally
  Interventions: Procedure: Repair of uterine incision; Procedure: Non exteriorization of the uterus

INTERVENTIONS:
Procedure: Repair of uterine incision
Procedure: Exteriorization of the uterus
  Arms: Exteriorization group
Procedure: Non exteriorization of the uterus
  Arms: Non exteriorization group

SUMMARY:
Cesarean section is one of the most frequently performed major operations worldwide. It accounts for between 1% and 70% of deliveries depending on the facilities or country assessed. In Egypt, the cesarean section rate is 22%, with higher rates seen in private hospitals. In 2015 ,incidence of cesarean section rate in Woman Health Hospital in Assiut university is 51.3% of all deliveries.

Different Operational techniques For cesarean section have been defined aimed at reducing surgical time, making the surgery easier and more efficient, lowering costs,decreasing the risk of adverse effects and postoperative morbidity, as well as length of hospital stay.

Also, Intraoperative blood loss is one of important complications during cesarean section. A systematic review included twenty one studies, in 2011, revealed that increase incidence of intraoperative blood loss and blood transfusion with increase number of cesarean deliveries.also anemia in the pregnancy increase maternal morbidities included intraoperative blood loss. In Egypt, prevalence of Iron deficiency anemia among pregnant women about 51% of pregnant women.

After baby born by cesarean section and the placenta has been extracted, uterine incision is sutured either by temporary removal of the uterus from the abdominal cavity (exteriorization of the uterus) to facilitate uterine incision repair or it is repaired within the abdominal cavity (in situ repair). There had been few randomized controlled trials comparing intraoperative and postoperative morbidity following exteriorization of the uterus with non-exteriorization. The conclusions drawn from these trials have been conflicting.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in 28 weeks
* Women who will undergo repeated lower segment cesarean section

Exclusion Criteria:

* First cesarean section
* Placenta previa.
* Rupture uterus.
* Classical caesarean section.(upper segment cesarean section)
* Sever Preeclampsia.
* Chorioamnionitis.
* prolonged or obstructed labour.
* Fibroid.
* Polyhydramnios.
* Multiple pregnancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1024 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss (mL) | 20 minutes
Postoperative Hemoglobin (gm/L) | 20 minutes

SECONDARY OUTCOMES:
Duration of operation (minutes) | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No